| The Effect of the Health Belief Model-Based Intervention in Primary School 3rd and 4th |
|---|
| Grade Students' Behavior on Safety Precautions for Preventing Accidents at School |
| NCT05576987 |
| Study Protocol and Statistical Analysis Plan |

June 3, 2022

## **Informed Consent Form**

The accidents causing deaths, temporary or permanent disabilities are a significant public health issue. In the 5-14 age group, injuries stand among the most critical causes of death and lifelong disabilities. Children in this age group spend a significant part of their day at school and are physically active within the school environment. This physical activity can lead to accidents and injuries. It is reported that 15% of child accidents occur at school. Therefore, it is important to enhance children's knowledge and behaviors regarding safety measures.

The aim of this study is to investigate the impact of a Health Belief Model-based intervention on the safety behaviors of 3rd and 4th-grade primary school students in school accidents.

Participants in the study will receive 30 minutes of training per week on school accidents for four weeks. Surveys will be conducted before and after the training to determine students' behaviors related to safety measures in school accidents. Participation is based on voluntary consent, and volunteers can withdraw from the study at any time.

Individual information will be kept confidential and will not be used for any other purpose. If you have any questions, you can contact the researcher whose name and phone number are provided below.

I have read the above information provided before the research. I have received written and verbal explanations about them. With these conditions, I give permission for my son/daughter to participate in the mentioned study.

Parent's Name, Signature, Date